CLINICAL TRIAL: NCT05196308
Title: Efficacy of Intracavernosal (Xeomin®) 100U as add-on Therapy to Sildenafil 100 mg on Demand Compared to Sildenafil 100 mg on Demand for the Treatment of Erectile Dysfunction (ED) Not Sufficiently Responsive to Standard Therapy With Phosphodiesterase Type 5 Inhibitors
Brief Title: Efficacy of Intracavernosal as add-on Therapy to Sildenafil 100 mg on Demand Compared to Sildenafil 100 mg on Demand for the Treatment of Erectile Dysfunction (ED) Not Sufficiently Responsive to Standard Therapy With Phosphodiesterase Type 5 Inhibitors
Acronym: MENOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP211042; 2021-005496-39 (EudraCT Number)
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; phosphodiesterase type 5 inhibitors; efficacy
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xeomin® receivers (Experimental): Patients will receive Xeomin®.
  Interventions: Drug: Investigational product administration Xeomin® (MERZ PHARMACEUTICALS GMBH)
- Placebo receivers (Placebo Comparator): Patients will receive placebo injection instead of Xeomin®.
  Interventions: Drug: Placebo administration

INTERVENTIONS:
Drug: Investigational product administration Xeomin® (MERZ PHARMACEUTICALS GMBH) — Administration of the investigational product.
  For the double-blind treatment phase, experimental group :
  Patients will receive Xeomin® (MERZ PHARMACEUTICALS GMBH), 100 U, a paired intracavernosal injection to be performed by the investigator.
  Arms: Xeomin® receivers
Drug: Placebo administration — For the double-blind treatment phase, control group :
  Patients will receive placebo of Xeomin® 100 U, a paired intracavernosal injection is to be performed by the investigator.
  Arms: Placebo receivers

SUMMARY:
The primary objective of this study is to investigate the efficacy of intracavernosal (Xeomin®) (100U) as add-on therapy to sildenafil 100 mg on demand in men with ED and insufficient response to standard therapy with 100 mg sildenafil on demand during the 4-week open-label run-in phase.

The secondary objectives are to further describe the efficacy and safety of (Xeomin®) 100U IC as add-on therapy to sildenafil 100 mg on demand:

1. to further assess efficacy using.

   * i) a log diary five-item questionnaire completed after each sexual attempt (Sexual Encounter Profile);
   * ii) a self-reporting measure that scores erection hardness on a 4 point scale completed after each sexual attempt;
   * iii) The Global Assessment Question.
2. to assess effect persistence at month 6 and month 9.
3. to assess safety of (Xeomin®) 100U IC in combination with sildenafil 100 mg on demand.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled study will be conducted in 9 centers, study participants will be adult men with ED and insufficient response to standard therapy with 100 mg sildenafil on demand during the 4-week open label run-in-phase, follow-up in the study will be 10±2 months.

This is a standard procedure to use placebo as control in studies assessing the efficacy of pharmacological treatment of ED. Furthermore the placebo group provides a benchmark for an objective analysis of safety and tolerability findings. The open-label run-in phase assures that only subjects who are true non-responders i.e. with insufficient response to standard therapy with 100 mg sildenafil prn during the 4-week open-label run-in phase are randomized and participate in the double-blind treatment phase.

Participants distributed between groups at a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

Subjects have to fulfill all of the following criteria before being included in the open-label run-in phase:

* Written informed consent obtained from the subject
* History of ED for at least 6 months prior to screening, defined as "the inability to achieve and maintain an erection of the penis sufficient to complete satisfactory sexual intercourse" (NIH), the diagnosis of ED has to be confirmed by a physician
* Understanding of study procedures and willingness to abide by all procedures during the course of the study
* Male subject aged ≥18 to ≤ 80 years at visit 1
* Have a monogamous relationship with a female sexual partner (vaginal penetration required for several of the primary efficacy variables) for at least 6 months prior to screening
* Highly motivated to obtain treatment for ED
* History of previous use of at least 1 marketed PDE5 inhibitor and insufficient therapeutic efficacy despite use of the highest approved dose

Subjects have to fulfill all of the following criteria before being included in the double blind treatment phase:

* At least 4 attempts at sexual intercourse during the open-label run-in phase with use of 100 mg sildenafil approximately 1 hour before attempting intercourse
* IIEF-EF score <17
* At least 50% of attempts at sexual intercourse during the open-label run-in phase had been unsuccessful i.e. the following question in the Subject Diary had to be answered with "No":

"Did your erection last long enough for you to have successful intercourse?" (SEP3: success in maintenance of erection)

* Highly motivated to obtain treatment for ED according to the investigator judgment
* Ability to understand and follow study-related instructions

Exclusion Criteria:

* Hypersensitivity to the active substance (Clostridium Botulinum neurotoxin type A) or to any of the excipients (Human albumin, sucrose)
* BW <50 kg
* ED caused by other primary sexual disorders including premature ejaculation or ED caused by untreated endocrine disease (eg, hypopituitarism, hypothyroidism, or hypogonadism)
* History of penile implant.
* The presence of clinically significant penile deformity in the opinion of the investigator.
* Patients with chronic stable angina treated with long-acting nitrates, or patients with chronic stable angina who have required short-acting nitrates in the last 90 days, or angina occurring during sexual intercourse in the last 6 months.
* Patients having met the criteria for unstable angina within 6 months prior to Visit 1, history of myocardial infarction or coronary artery bypass graft surgery within 90 days prior to Visit 1, or percutaneous coronary intervention (eg, angioplasty or stent placement) within 90 days prior to Visit 1.
* Any supraventricular arrhythmia with an uncontrolled ventricular response (mean heart rate >100 bpm) at rest despite medical or device therapy, or any history of spontaneous or induced sustained ventricular tachycardia (heart rate >100 bpm for 30 sec) despite medical or device therapy, or the presence of an automatic internal cardioverter-defibrillator.
* A history of sudden cardiac death (arrest) despite medical or device therapy.
* Any evidence of congestive heart failure within 6 months prior to Visit 1.
* A significant conduction defect within 90 days prior to Visit 1.
* Systolic blood pressure >170 or <90 mm Hg or diastolic blood pressure >100 or <50 mm Hg at screening (if stress is suspected, retest under basal conditions), or patients with malignant hypertension.
* <12 weeks since most recent injection of BTX-A/B into any body region for any indication
* Neurological disorder associated with neuro muscular dysfunction of any kind in medical history.
* Planned concomitant treatment with BTX -A/B of any body region during the study.
* Known hypersensitivity to human serum albumin, sucrose, or the active substance BTX-A.
* Generalized disorders of muscles activity (e.g. myasthenia gravis, Lambert-Eaton-Syndrome, amyotrophic lateral sclerosis) or any other significant peripheral neuromuscular dysfunction which might interfere with the study.
* Any condition that would interfere with the patient's ability to provide informed consent or comply with study instructions, would place patient at increased risk, or might confound the interpretation of the study results.
* Current treatment with nitrates (as outlined in previous Exclusion Criterion, cancer chemotherapy, or anti-androgens.
* History of drug, alcohol, or substance abuse within the past 6 months.
* Investigators, site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
* Treatment within the last 30 days with a drug or device that has not received regulatory approval at the time of study entry.
* Ongoing severe or uncontrolled systemic disease, current malignancy, haemophilia, or HIV infection in medical history.
* Severe or uncontrolled respiratory disease in medical history.
* Evidence or suspicion that the subject is not willing or unable (e.g.due to severe cognitive communication impairment) to understand the information that is given to him as part of the informed consent, in particular regarding the risks and discomfort which he would agree to be exposed to.
* Any reason which in the investigator's opinion is likely to compromise the subject's ability to participate in the study.
* Subject who is imprisoned or is lawfully kept in an institution
* Participation in a clinical study within 12 weeks prior to screening or planned participation during this study.
* Previous participation in this clinical study.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male subject aged ≥18 to ≤ 80 years at visit1
Enrollment: 226 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Change in the erectile function | at baseline and month 3
  Change in the erectile function between baseline and month 3, measured by the International Index of Erectile Function - Erectile Function domain score (IIEF-EF).
  The International Index of Erectile Function (IIEF) is a 15-item self-report instrument assessing male sexual function. The Erectile Function (EF) domain score of the IIEF, comprised of items 1 to 5 and 15 from the IIEF, is used in this study.
Change in SEP2 | at baseline and month 3
  Question providing information as whether the erection is hard enough to penetrate (SEP2).
  The SEP is a log diary with 5 questions answered after each sexual intercourse attempt, providing information as to whether the erection was hard enough to penetrate (SEP 2), or whether it was maintained for completion (SEP 3) or a satisfactory sexual experience (SEP 4).
Change in SEP3 | at baseline and month 3
  Question providing information as duration of erectile.
  The SEP is a log diary with 5 questions answered after each sexual intercourse attempt, providing information as to whether the erection was hard enough to penetrate (SEP 2), or whether it was maintained for completion (SEP 3) or a satisfactory sexual experience (SEP 4).

SECONDARY OUTCOMES:
Change in SEP 4 score | at baseline and month 3
  Percentage of SEP 4 of the Sexual Encounter Profile questionnaire
  The SEP is a log diary with 5 questions answered after each sexual intercourse attempt, providing information as to whether the erection was hard enough to penetrate (SEP 2), or whether it was maintained for completion (SEP 3) or a satisfactory sexual experience (SEP 4).
The Erection Hardness Score (EHS) | at baseline and month 3
  Change in the mean Erection Hardness Score at 3-, month (±2 weeks) after placebo or Xeomin® 100U IC injection compared to baseline. (Mulhall JP et al. Validation of the erection hardness score. J Sex Med. 2007;4(6):1626-1634). The EHS is a single-item Likert scale. The tool asks men to consider the question 'How would you rate the hardness of your erection?' and select one of the options below:
  0 - Penis does not enlarge; 1 - Penis is larger, but not hard; 2 - Penis is hard, but not hard enough for penetration; 3 - Penis is hard enough for penetration, but not completely hard; 4 - Penis is completely hard and fully rigid.
Global Assessment Question (GAQ) | at baseline and month 3
  "Has the treatment you have been taking over the past 4 weeks improved your erections? (Please compare your current erections after treatment with your erections before your participation in this study)": yes or no: Change in the percentage of "yes" answer at 3-month (±2 weeks) after placebo or Xeomin® 100U IC injection compared with baseline.
Persistence of efficacy | at 6- and 9- month
  Persistence of efficacy at 6- and 9- month post-treatment administration using the same tools (IIEF-EF, SEP, EHS, GAQ) among patients for whom treatment has been assessed as efficient individually.
  Individual efficacy of treatment in each patient will be assessed using minimally clinically important difference (MCID) for the IIEF-EF domain according to ED severity (Rosen 2011) i. e. MCID ≥ 5 for moderate ED (IIEF-EF 11-16) and MCID ≥ 7 for severe ED (IIEF-EF6-10).

CONTACTS AND LOCATIONS:
Overall Officials: François GIULIANO, MD, PhD, Principal Investigator — Neuro-Urology-Andrology, Raymond Poincaré Hospital, APHP
Locations (1):
- Neuro-Urology-Andrology, Physical Medicine and Rehabilitation Department, Raymond Poincaré Hospital, APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher WA, Gruenwald I, Jannini EA, Lev-Sagie A, Lowenstein L, Pyke RE, Reisman Y, Revicki DA, Rubio-Aurioles E. Standards for Clinical Trials in Male and Female Sexual Dysfunction: III. Unique Aspects of Clinical Trials in Male Sexual Dysfunction. J Sex Med. 2017 Jan;14(1):3-18. doi: 10.1016/j.jsxm.2016.08.016. PMID 28065358
- [Background] Mulhall JP, Goldstein I, Bushmakin AG, Cappelleri JC, Hvidsten K. Validation of the erection hardness score. J Sex Med. 2007 Nov;4(6):1626-34. doi: 10.1111/j.1743-6109.2007.00600.x. Epub 2007 Sep 21. PMID 17888069
- [Derived] Giuliano F, Denys P, Joussain C. Effectiveness and Safety of Intracavernosal IncobotulinumtoxinA (Xeomin(R)) 100 U as an Add-on Therapy to Standard Pharmacological Treatment for Difficult-to-Treat Erectile Dysfunction: A Case Series. Toxins (Basel). 2022 Apr 16;14(4):286. doi: 10.3390/toxins14040286. PMID 35448895